CLINICAL TRIAL: NCT02873923
Title: Survival Endpoints in Randomized Clinical Trials in Sarcoma Patients: Meta-analyses for the Assessment of the Impact Various Definitions on Trials' Results and of Surrogate Properties for OS
Brief Title: Variability of Definitions for Survival Endpoints and Surrogate Properties for OS in Sarcoma Trials: a Meta-analysis
Acronym: DATECAN-2
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: IB2012-DATECAN-2
Record Dates: First submitted 2016-08-09; First posted 2016-08-22 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-12

CONDITIONS: Cancer
Keywords: clinical trial; surrogate endpoints; meta analysis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a metastatic soft tissue sarcoma: All patients included in eligible clinical trials of the meta-analysis
  Interventions: Drug: undefined

INTERVENTIONS:
Drug: undefined — Chemotherapy drug (meta-analyses of randomized trials)

SUMMARY:
The DATECAN-2 project aims at assessing the surrogate properties for OS of several time-to-event endpoints through meta-analyses of completed and published randomized controlled trials. Two main cancer localization are concerned: breast cancer and soft-tissue sarcomas. The impact of survival endpoints' definitions on the trials' results and conclusions will also be evaluated.

DETAILED DESCRIPTION:
Background: In randomized phase III cancer clinical trials, the validated and most objectively defined evaluation criterion is overall survival (OS). Therapeutic progress, which in certain contexts has significantly reduced overall mortality, the development of new types of cytostatic treatments (as opposed to cytotoxic treatments), the current context of strategic trials and the multiplication of lines of treatment have resulted in the necessity of creating new evaluation criteria measuring treatment efficacy sooner and more precisely: for example, progression-free survival in second line treatment, duration of local control, and time until treatment failure. These types of surrogate endpoints are commonly used in phase II trials but are increasingly being used to replace overall survival in phase III trials. Their development is strongly influenced by the necessity of reducing clinical trial duration, cost and number of patients.

However while these survival endpoints are frequently used, they are often poorly defined and when they are, the definition can vary between trials. The lack of standardized definitions constitutes a clear limitation to their use as primary endpoints. Furthermore, this variability of definitions can have an important impact on trials' results by affecting power and estimation.

The ongoing DATECAN-1 project is aimed at providing guidelines for the definitions of survival endpoints in cancer trials (2009-2011 grant from the French League Against Cancer). Standardized recommendations will be available for survival endpoints commonly used for various cancer sites including pancreas, sarcomas and GIST (gastro-intestinal stromal tumors), breast, stomach.

Objectives: Following these guidelines, one can wonder how sensitive are these definitions? Or similarly, how do survival endpoints' definitions impact the conclusions of clinical trials? The objective of the DATECAN-2 study is to assess the impact of survival endpoints' definitions, as defined by the consensus guidelines, on trials' results and conclusions. The second objective is to study the surrogate properties for OS of these survival endpoints.

Methods: The evaluation of the impact of the variability of the definitions of survival endpoints on the results of clinical trials will be evaluated using individual data from datasets collected in the context of published (academic) clinical trials, as well as simulated datasets.

After approval by the sponsors, data will be analyzed using various endpoints' definitions including (i) the definition provided in the publication and (ii) the definition provided by the guidelines. We will identify which survival endpoint, as defined by the guidelines, was reported in the publication. Next, realistic data sets will be simulated that mimic data that could be observed in randomized cancer trials. We will generate data sets with varying proportions of events (number of deaths, progression, etc) depending on the survival endpoints of interest. Survival endpoints will be compared across treatment arms using the definition provided by the guidelines, and based on various scenarios (different proportions of events, length of follow-up, etc).

Using data from published data sets, we will evaluate survival endpoints in terms of surrogate candidates for OS. A hierarchy of the survival endpoints will be proposed according to their surrogate properties based on two criteria: the Fleming classification and the R2 value for validated surrogates. Depending on the number of clinical trials, single-trial or multiple-trials method will be employed. Single-trial methodology relies on Prentice criteria and Freedman's proportion of treatment effect (PTE) explained by the surrogate. In case of multiple trials, and when meta-analysis of clinical trials is feasible, surrogacy of candidate endpoints for OS will also be explored using weighted linear regression, which jointly estimates the level of association between endpoints and the trial-level association (R²) between treatment effects on the candidate surrogate and the final endpoint. Based on these results (R² and PTE), survival endpoints will be ranked according to their surrogate capabilities for OS.

Expected results: Analysis of the sensitivity of clinical trials' results to the survival endpoints' definitions and surrogacy properties are key features when designing and conducting clinical trials. Based on our results, we will be able to anticipate the expected impact of the definitions on effect size, sample size and power. We will be able to estimate these parameters more precisely and as such provide more efficient estimations. Similarly our assessment of the surrogate properties of the survival endpoints should help us for the selection of the best surrogate marker for OS, and thus limit biases. Overall, by producing less biased results and more efficient designs, our project should have an important role in the design and conduct of future randomized trials.

ELIGIBILITY:
No patient will be included.

This project concern Phase III clinical trials with following criteria :

Inclusion Criteria:

* Phase III clinical trials that included overall survival (OS) as endpoint and another time-to-event endpoint as primary or secondary endpoint
* Phase III clinical trials that included patients with metastatic soft tissue sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in phase III randomized clinical trials assessing patients with metastatic soft-tissue sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 2846 (Actual)
Dates: Start 2012-10; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Savina M, Gourgou S, Italiano A, Dinart D, Rondeau V, Penel N, Mathoulin-Pelissier S, Bellera C. Meta-analyses evaluating surrogate endpoints for overall survival in cancer randomized trials: A critical review. Crit Rev Oncol Hematol. 2018 Mar;123:21-41. doi: 10.1016/j.critrevonc.2017.11.014. Epub 2017 Nov 23. PMID 29482777
- [Result] Savina M, Litiere S, Italiano A, Burzykowski T, Bonnetain F, Gourgou S, Rondeau V, Blay JY, Cousin S, Duffaud F, Gelderblom H, Gronchi A, Judson I, Le Cesne A, Lorigan P, Maurel J, van der Graaf W, Verweij J, Mathoulin-Pelissier S, Bellera C. Surrogate endpoints in advanced sarcoma trials: a meta-analysis. Oncotarget. 2018 Oct 2;9(77):34617-34627. doi: 10.18632/oncotarget.26166. eCollection 2018 Oct 2. PMID 30349653

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
Started | 2846
Completed | 2846
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
Number analyzed (Participants) | 2846
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2846
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1423
  Male | 1423

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of deaths
Time Frame: up to 18 months following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
Number analyzed (Participants) | 2846
Participants | 1704

2. Secondary Outcome: Progression-free Survival
Description: Number of progressions or deaths. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 12 months following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
Number analyzed (Participants) | 2846
Participants | 2303

3. Post Hoc Outcome: Individual-level Association
Description: Individual-level association between 12-month progression-free survival and 18-month overall survival
Time Frame: within 18 months following randomization
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
Number analyzed (Participants) | 2846
Correlation coefficient | 0.66 [0.63 to 0.68]
Statistical Analysis 1: Comparison: Patients With a Metastatic Soft Tissue Sarcoma; Test type: Other; Correlation coefficient = 0.66, 95% CI 2-sided [0.63 to 0.68]; As of today, the meta-analytic surrogacy evaluation scheme proposed by Buyse and Burzykowski et al. is considered as the most statistically rigorous method for the validation of surrogate endpoints. This approach requires individual-patient data (IPD) from multiple randomized clinical trials (RCT) with similar design and treatment to address surrogacy from a multi-level framework. At the patient level, the surrogate endpoint should be correlated and predictive of the final endpoint regardless of the treatment (individual level association). At the trial level, the treatment effect on the surrogate endpoint should be correlated and predictive of the treatment effect on the final endpoint (trial-level association). Individual-level and trial-level associations estimated using weighted linear regression and the two-stage model introduced by Buyse and Burzykowski

4. Post Hoc Outcome: Trial-level Association
Description: Trial-level association between 12-month progression-free survival and 18-month overall survival
Time Frame: within 18 months following randomization
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
Number analyzed (Participants) | 2846
Correlation coefficient | 0.00 [0.00 to 0.05]
Statistical Analysis 1: Comparison: Patients With a Metastatic Soft Tissue Sarcoma; Test type: Other; correlation coefficient = 0.00, 95% CI 2-sided [0.00 to 0.005]; [other analysis details as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 18 months following randomization
Description: This study is a meta-analysis focussing on the association between progression-free survival and overall survival. As such, we did not report on the safety.
  Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Patients With a Metastatic Soft Tissue Sarcoma
All-Cause Mortality (participants affected / at risk) | 1704/2846
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes